CLINICAL TRIAL: NCT02382731
Title: Interventions to Support Long-Term Adherence aNd Decrease Cardiovascular Events Post-Myocardial Infarction
Acronym: ISLAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: #06683
Record Dates: First submitted 2015-03-02; First posted 2015-03-09 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Myocardial Infarction; Coronary Disease
MeSH Terms: conditions — Myocardial Infarction; Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual care (No Intervention): Usual care (no intervention)
- Usual care + letters (Experimental): Usual care plus a series of postal educational reminders (including information for patients to share with clinicians)
  Interventions: Behavioral: Usual care + letters
- Usual care + letters + automated calls (Experimental): Usual care plus a series of postal educational reminders (including information for patients to share with clinicians), plus automated reminder interactive voice response phone calls to identify patients at being at risk for non-adherence and a trained lay health worker to provide additional support and navigation for such patients via telephone.
  Interventions: Behavioral: Usual care + letters + automated calls

INTERVENTIONS:
Behavioral: Usual care + letters — A series of five postal educational reminders sent on behalf of each hospital's interventional cardiology team to the patient approximately 4, 8, 20, 32, and 44 weeks post-MI procedure, with an insert for the family physician and pharmacist at approximately 4 and 8 weeks post-MI procedure.
  Arms: Usual care + letters
Behavioral: Usual care + letters + automated calls — A series of five postal educational reminders as per the usual care + letters arm plus interactive voice response phone calls to the patient delivered approximately 2 weeks after the letters, as well as personalized telephone follow up by trained lay health workers for patients identified by the interactive voice response system as non-adherent. The automated algorithm is designed to identify patients who are non-adherent and who may benefit from personalized educational phone call and/or system navigation support by the lay health worker. Lay health workers will not provide clinical advice.
  Arms: Usual care + letters + automated calls

SUMMARY:
Proven treatments exist that improve quality of life and reduce the risk of repeat heart attacks or death amongst persons who have already had one heart attack. These treatments include medications and supervised cardiac rehabilitation programs. Unfortunately, research shows that many people who have had a heart attack do not stick with these treatments and therefore cannot benefit. This quality improvement research program seeks to understand the impact of interventions that could be readily implemented at scale by entire health systems or organizations wishing to improve adherence to proven treatments. Specifically, the trial will test whether providing Ontario-based patients (and their health professionals) with repeated educational reminders delivered via post and phone will help improve the use of medications or attendance at cardiac rehabilitation. During the project, the types of patients who are most responsive will be identified as will the most cost-effective strategy for delivering reminders. The trial team are partnering in this project with health system decision makers who have an interest in using the results to create standard operating procedures that could benefit patients across the province.

DETAILED DESCRIPTION:
EXECUTIVE SUMMARY

Background: In patients who have had a myocardial infarction (MI) and coronary disease, guidelines recommend cardiac rehabilitation services and the long-term use of cardiac medications to reduce the risk of recurrent cardiovascular events. Adherence to these recommendations substantially reduces morbidity and mortality post-MI. However, for a variety of patient, provider, and system-level reasons, adherence to cardiac medications declines to approximately 50% by 12 months. Likewise, only 30-40% of patients participate in cardiac rehabilitation. Thus, interventions to increase secondary prevention treatment adherence are urgently needed.

The Cardiac Care Network of Ontario (CCN) holds a registry of all patients in the province who have a coronary angiography. The registry has been used to identify gaps in care and to plan health system strategies for high-risk patients. More recently, a pilot trial was conducted in Hamilton by the trial team using data in the registry to send recurrent postal reminders regarding the importance of treatment adherence to patients, their pharmacists, and family physicians. A similar program is underway in Ottawa using automated phone calls with interactive voice response and nurse follow up. These interventions both have the potential to address known determinants of adherence. The CCN, Ministry of Health and Long-Term Care, Health Quality Ontario, and other stakeholders across Ontario are interested in evaluating the comparative effectiveness and costs of these interventions.

Research Questions: The research objectives were formed by the decision makers' need to evaluate whether and in what format to sustain and/or scale-up post-MI educational reminder interventions:

i. Can educational reminders delivered via post and/or using interactive voice response with personalized telephone follow up improve secondary prevention treatment adherence post-MI?

ii. How do different approaches to improve adherence to these recommendations compare in terms of clinical effectiveness and costs?

iii. Which subgroups are more/less likely to respond to reminders?

Research Approach: This is a pragmatic, randomized controlled trial with blinded outcome assessment. Patients in cardiac centres throughout Ontario who undergo a coronary angiography will be provided a letter of information explaining the study appended to the standard CCN letter of information. CCN will identify eligible patients (those with substantial coronary artery disease who survive their initial hospitalization post-MI) and provide the patient list back to the cardiac centre. A representative at the centre will securely send this list to the Population Health Research Institute in Hamilton. Patients will be randomized by the Population Health Research Institute team to one of three arms:

1. - Usual care, with no standardized educational materials or reminders
2. - Postal letters sent from Population Health Research Institute on behalf of each hospital's interventional cardiology team to the patient approximately 4, 8, 20, 32, and 44 weeks post-MI, with an insert for the family physician and pharmacist at approximately 4 and 8 weeks post-MI.
3. - Postal letters as above plus interactive voice response phone calls to the patient delivered approximately 2 weeks after the letters, as well as personalized telephone follow up by trained lay health workers for patients identified by the interactive voice response system as non-adherent.

Patient self-report and administrative data will be used to assess outcomes 12 months post-MI. Analyses will be by intention to treat. The primary outcome is adherence to guideline-recommended treatments. Secondary outcomes include health services utilization (including outpatient visits to interventional cardiology), recurrent cardiovascular events, and mortality. During the trial, a theory-informed process questionnaire will be administered to a random sub-sample. An economic evaluation will be conducted from the perspective of the public health care payer.

Implications: This project has the potential to lead to improvements in care for patients at high cardiovascular risk as well as provide generalizable insights regarding how to optimize interventions to improve adherence. Further, it has the potential to inform how other health databases could be used to improve health system performance.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older having a coronary angiography following a myocardial infarction (ST-elevation myocardial infarction or non-ST-elevation myocardial infarction), with evidence of coronary artery disease (>50% blockage of left main or >70% blockage of ≥1 major cardiac arteries).
* Discharged from the catheterization centre alive, either home or to a local (non-cardiac) hospital
* Patients must be Ontario residents

Exclusion Criteria:

* Patients will be excluded if they expire during their hospitalization or if they have cardiogenic shock (Killip Class 4) at the time of their post-MI coronary angiography due to their poor prognosis.(El-Menyar et al., 2012)
* Patients will also be excluded if they require a translator to receive services in English as recorded in the CCN referral form, as it is infeasible to offer the interventions in multiple languages at this stage.
* Patients whose data are not complete and received in time to deliver the first post-procedure intervention will be excluded as they cannot receive the intervention as intended.
* Patients who do not have an Ontario health card number

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2742 (Actual)
Dates: Start 2015-09; Primary Completion 2017-06 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Medication adherence | 12 months post-MI
  Number of cardiac medication classes with no missed tablets in last week (ordinal) [patient report]
Cardiac rehabilitation completion | 12 months post-MI
  Patient attended at least one of the rehabilitation components and formal re-assessment at the conclusion of the program (dichotomous) [patient report]

SECONDARY OUTCOMES:
Cardiac rehabilitation attendance | 12 months post-MI
  Participation, defined as attending at least one exercise session following enrolment assessment (dichotomous) [patient report]
Quality of life | 12 months post-MI
  Seattle Angina Questionnaire-7 [patient report]
Treatment discussion | 12 months post-MI
  Adherence to both medication and exercise discussed with providers in last three months (dichotomous) [patient report]
Smoking status | 12 months post-MI
  Point-prevalence, smoking any cigarettes in last three months (dichotomous) [patient report]
Medication persistence | 12 months post-MI
  Active prescription for ALL recommended medications (dichotomous) [patient report]
Medication persistence | 12 months post-MI
  Active prescription for EACH recommended medication (dichotomous) [patient report]
Medication adherence | 12 months post-MI
  No missed tablets in last week for ANY recommended medication (dichotomous) [patient report]
Medication adherence | 12 months post-MI
  No missed tablets in last month for any recommended medication (dichotomous)[patient report]
Medication adherence | 12 months post-MI
  No missed tablets in last month for ANY recommended medication (dichotomous) [patient report]
Medication adherence | 12 months post-MI
  Number of missed tablets in last week for EACH recommended medication (continuous, 0 to 28) [patient report]
Medication adherence | 12 months post-MI
  Number of missed tablets in last month for each recommended medication (continuous, 0 to 28) [patient report]
Medication adherence | 12 months post-MI
  Medication possession ratio > 80% for ALL recommended medications in those 65+ (dichotomous) [administrative data]
Medication adherence | 12 months post-MI
  Medication possession ratio > 80% for EACH of the recommended medications in those 65+ (dichotomous) [administrative data]
Medication adherence | 12 months post-MI
  Mean medication possession ratio for ALL recommended medications in those 65+ (continuous, 0 to 100) [administrative data]
Medication adherence | 12 months post-MI
  Mean medication possession ratio for EACH recommended medication in those 65+ (continuous, 0 to 100) [administrative data]
Cardiovascular event | 12 months post-MI
  Coronary bypass surgery or stent or repeat MI (dichotomous) [administrative data]
Mortality | 12 months post-MI
  Death during follow-up [administrative data]
Health utilization | 12 months post-MI
  Outpatient visits (count) [administrative data]
Health utilization | 12 months post-MI
  Emergency Room visits not leading to admission (count) [administrative data]
Health utilization | 12 months post-MI
  Hospitalizations (count) [administrative data]

CONTACTS AND LOCATIONS:
Overall Officials: Noah Ivers, Principal Investigator — Women's College Hospital; John-David Schwalm, Principal Investigator — Population Health Research Institute; Madhu Natarajan, Principal Investigator — Population Health Research Institute; Jeremy Grimshaw, Principal Investigator — Ottawa Hospital Research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Menyar A, Zubaid M, AlMahmeed W, Sulaiman K, AlNabti A, Singh R, Al Suwaidi J. Killip classification in patients with acute coronary syndrome: insight from a multicenter registry. Am J Emerg Med. 2012 Jan;30(1):97-103. doi: 10.1016/j.ajem.2010.10.011. Epub 2010 Dec 14. PMID 21159479
- [Derived] McCleary N, Ivers NM, Schwalm JD, Witteman HO, Taljaard M, Desveaux L, Bouck Z, Grace SL, Grimshaw JM, Presseau J. Impacts of two behavior change interventions on determinants of medication adherence: process evaluation applying the health action process approach and habit theory alongside a randomized controlled trial. J Behav Med. 2022 Oct;45(5):659-673. doi: 10.1007/s10865-022-00327-0. Epub 2022 May 20. PMID 35596020
- [Derived] Desveaux L, Saragosa M, Russell K, McCleary N, Presseau J, Witteman HO, Schwalm JD, Ivers NM. How and why a multifaceted intervention to improve adherence post-MI worked for some (and could work better for others): an outcome-driven qualitative process evaluation. BMJ Open. 2020 Sep 3;10(9):e036750. doi: 10.1136/bmjopen-2019-036750. PMID 32883724
- [Derived] Ivers NM, Schwalm JD, Bouck Z, McCready T, Taljaard M, Grace SL, Cunningham J, Bosiak B, Presseau J, Witteman HO, Suskin N, Wijeysundera HC, Atzema C, Bhatia RS, Natarajan M, Grimshaw JM. Interventions supporting long term adherence and decreasing cardiovascular events after myocardial infarction (ISLAND): pragmatic randomised controlled trial. BMJ. 2020 Jun 10;369:m1731. doi: 10.1136/bmj.m1731. PMID 32522811